CLINICAL TRIAL: NCT00142012
Title: School-Based Obesity Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of Pennsylvania (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-OPHR-321534
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2005-11-17 (Estimated); Status verified 2005-09

CONDITIONS: Obesity
Keywords: School-based; Obesity; Prevention
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

INTERVENTIONS:
Behavioral: Nutrition Intervention

SUMMARY:
The overarching goal of this initiative is to reduce the prevalence and occurrence of obesity and increase the remission of obesity in children and adolescents through implementation of a Comprehensive School Nutrition Policy designed to promote changes in the school environment that will reinforce students' development of healthy eating and physical activity patterns inside and outside of school.

DETAILED DESCRIPTION:
The proposed research aims to evaluate the effects of a school-based nutrition policy initiative on prevalence, incidence and remission of overweight (BMI > 95th percentile). It is a partnership between the Food Trust, the School District of Philadelphia and the University of Pennsylvania. Participants are approximately 1500 students from ten schools in grades four through eight. Half of the schools were randomized to a comprehensive School Nutrition Policy Initiative (SNPI) based on CDC's Guidelines to Promote Lifelong Healthy Eating. The SNPI is a community-based intervention administered by the Comprehensive School Nutrition Policy Task Force that is comprised of 40 individuals representing the public and private sectors. The goal of the SNPI is to change the school environment to: support healthy eating, increase physical activity, and decrease the prevalence of childhood overweight and diet-related diseases. The remaining study participants are in five control schools, matched for ethnicity, SES, and type of food service. Most students are African American and qualify for free and reduced meals at school (household income < 185% of the poverty level adjusted for household size). Assessments of weight, height, intake, activity, inactivity and eating disorder symptomatology are being conducted at baseline and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Any child in 4th, 5th, 6th grades in study site schools

Exclusion Criteria:

* Any child not in 4th, 5th, 6th in study site schools

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500
Dates: Start 2002-10; Study Completion 2005-06

PRIMARY OUTCOMES:
Weightloss
Weight maintenance

SECONDARY OUTCOMES:
Risk for overweight status (BMI 85th to 95th percentile)
BMI z-scores, calculated for a given age and gender, will show a greater decline in intervention subjects versus controls

CONTACTS AND LOCATIONS:
Overall Officials: Gary D. Foster, PhD, Principal Investigator — U. of Pennsylvania